CLINICAL TRIAL: NCT05611736
Title: Effects of Intracanal Cryotherapy on Postoperative Pain in Necrotic Teeth With Symptomatic Apical Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Effects of Intracanal Cryotherapy on Endodontic Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Muhammad Zubair Ahmad, Associate Professor, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-19-08
Record Dates: First submitted 2022-10-28; First posted 2022-11-10 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Dental Pulp Necroses; Apical Periodontitis; Post Operative Pain
Keywords: Cryotherapy; endodontic pain; molar teeth; root canal treatment
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis; Pain, Postoperative | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cold saline (Experimental): After standard chemo-mechanical preparation of the root canal, final irrigation will be performed using 20 milliliters of cold (at 2.5 degrees Celsius temperature) saline solution.
  Interventions: Other: cold saline
- saline (Active Comparator): After standard chemo-mechanical preparation of the root canal, final irrigation of the root canal system will be performed using 20 milliliters of normal saline solution at room temperature.
  Interventions: Other: saline

INTERVENTIONS:
Other: cold saline — After standard chemo-mechanical preparation of the root canal, final irrigation will be performed using 20 milliliters of cold (at 2.5 degrees Celsius temperature) saline solution.
  Other Names: cold normal saline
  Arms: cold saline
Other: saline — After standard chemo-mechanical preparation of the root canal, final irrigation of the root canal will be done using normal saline solution at room temperature
  Other Names: normal saline
  Arms: saline

SUMMARY:
The goal of this clinical trial is to evaluate the effect of cold saline (2.5 degrees Celsius) irrigation on postoperative pain in patients who require root canal treatment in molar teeth because of dead dental pulp and infection around the apex of the root of the involved teeth. This cold saline irrigation will be done after standard irrigation of the canal using a 5.25% sodium hypochlorite solution. The main questions it aims to answer are:

* Is there any difference in postoperative pain when final irrigation is performed using a cold saline solution compared to the irrigation using the saline solution at room temperature in patients who require dental root canal treatment of molar teeth?
* Because of cold saline irrigation, what type of adverse event/s may result?

Participants will be asked to fill out a questionnaire before the start of the root canal treatment and record the preoperative pain using the visual analog scale (VAS). Root canal treatment will be completed in one visit. The standard procedure of root canal treatment will be followed, including irrigation of the canal using 5.25% sodium hypochlorite. As a final irrigation, either cold saline solution or a normal saline solution at room temperature will be used. The participants will be asked to fill out another questionnaire and record the presence, duration, and intensity of postoperative pain, and if painkiller medicine was taken immediately after completion of root canal treatment and at 6 hours, 12 hours, 72 hours, and 1-week intervals.

The researcher will compare the effect of the final irrigation of a cold saline solution with that of a normal saline solution at room temperature on postoperative pain.

DETAILED DESCRIPTION:
Postoperative pain in root canal therapy is multifactorial in nature, including changes in periapical pressure, microbial factors, inflammatory mediators, and psychological factors. Postoperative pain in endodontics between visits or after completion of the treatment is a major concern to both patients and operators. Teeth presented with preoperative pain, irreversible pulpitis, pulp necrosis, and apical periodontitis are the most susceptible to postoperative pain The pharmacological management of pain using medications such as nonsteroidal anti-inflammatory drugs, paracetamol, or corticosteroids, despite being relatively safe, can have side effects such as gastrointestinal intolerance and renal, hepatic, and respiratory disorders such as asthma which have been reported in the literature. To avoid these secondary effects, intracanal medications, laser, and cryotherapy have been suggested in the literature.

Physical and clinical evidence suggests that the application of cold may decrease pain through the mechanism of decreasing the conduction velocity of nerve signals, hemorrhage, edema, and local inflammation. An in vitro study showed that intracanal irrigation with cold saline at 2.5 degrees Celsius reduced the external root surface temperature by more than 10 degrees Celsius, which would be enough to produce the anti-inflammatory effect in peri-radicular tissues.

There are very few studies done to evaluate the effect of intracanal cryotherapy on postoperative pain in root canal therapy.

This clinical trial aims to assess if final irrigation using cold saline solution after standard chemo-mechanical preparation (root canal instrumentation and irrigation using 5.25% sodium hypochlorite) procedures results in any difference in the incidence and intensity of postoperative pain in patients presenting with molar teeth with necrosis of pulp and symptomatic apical periodontitis. This clinical trial will also assess the incidence of any adverse event as a result of cold saline irrigation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* Patients with maxillary or mandibular molar teeth that require root canal treatment
* The diagnosis of pulp necrosis
* The presence of symptomatic apical periodontitis
* The presence of normal occlusion

Exclusion Criteria:

* Previously done root canal treatment
* Pregnancy
* Presence of any systemic disease or allergic reactions
* Use of any analgesic or antibiotic medications within the past three days
* Sinus tract or local gingival swelling around the affected tooth
* Periodontal pocket greater than 3 mm around the affected tooth
* Severe periodontal disease
* Internal or external root resorption
* Broken files
* Over instrumentation
* Incomplete filling of the root canal
* Overfilling of the root canal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 6 hours postoperatively
  Postoperative pain will be measured using visual analog scale (VAS)
Postoperative pain | 24 hours postoperatively
  Postoperative pain will be measured using visual analog scale (VAS)
Postoperative pain | 72 hours postoperatively
  Postoperative pain will be measured using visual analog scale (VAS)
Postoperative pain | 1 week postoperatively
  Postoperative pain will be measured using visual analog scale (VAS)
adverse event | during the irrigation procedure
  If any adverse event will occur, it will be recorded
adverse event | immediately after the irrigation procedure
  If any adverse event will occur, it will be recorded
adverse event | 6 hours postoperatively
  If any adverse event will occur, it will be recorded
adverse event | 24 hours postoperatively
  If any adverse event will occur, it will be recorded
adverse event | 72 hours postoperatively
  If any adverse event will occur, it will be recorded
adverse event | 1 week postoperatively
  If any adverse event will occur, it will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Zubair Ahmad, BDS, FCPS, Principal Investigator — Qassim University
Locations (1):
- Muhammad Zubair Ahmad, Ar Rass, Al-Qassim Region, Saudi Arabia

REFERENCES:
- [Background] Vera J, Ochoa-Rivera J, Vazquez-Carcano M, Romero M, Arias A, Sleiman P. Effect of Intracanal Cryotherapy on Reducing Root Surface Temperature. J Endod. 2015 Nov;41(11):1884-7. doi: 10.1016/j.joen.2015.08.009. Epub 2015 Oct 1. PMID 26433855
- [Background] Alharthi AA, Aljoudi MH, Almaliki MN, Almalki MA, Sunbul MA. Effect of intra-canal cryotherapy on post-endodontic pain in single-visit RCT: A randomized controlled trial. Saudi Dent J. 2019 Jul;31(3):330-335. doi: 10.1016/j.sdentj.2019.03.004. Epub 2019 Mar 14. PMID 31337936
- [Background] Fayyad DM, Abdelsalam N, Hashem N. Cryotherapy: A New Paradigm of Treatment in Endodontics. J Endod. 2020 Jul;46(7):936-942. doi: 10.1016/j.joen.2020.03.019. Epub 2020 May 6. PMID 32386857
- [Background] Sadaf D. Limited Quality Evidence Suggests that Application of Cryotherapy May Be Helpful in Reducing Postoperative Pain in Root Canal Therapy in Patients With Symptomatic Apical Periodontitis. J Evid Based Dent Pract. 2019 Jun;19(2):195-197. doi: 10.1016/j.jebdp.2019.05.005. Epub 2019 May 6. PMID 31326055
- [Background] Gundogdu EC, Arslan H. Effects of Various Cryotherapy Applications on Postoperative Pain in Molar Teeth with Symptomatic Apical Periodontitis: A Preliminary Randomized Prospective Clinical Trial. J Endod. 2018 Mar;44(3):349-354. doi: 10.1016/j.joen.2017.11.002. Epub 2018 Feb 3. PMID 29398090
- [Background] Sadaf D, Ahmad MZ, Onakpoya IJ. Effectiveness of Intracanal Cryotherapy in Root Canal Therapy: A Systematic Review and Meta-analysis of Randomized Clinical Trials. J Endod. 2020 Dec;46(12):1811-1823.e1. doi: 10.1016/j.joen.2020.08.022. Epub 2020 Sep 8. PMID 32916207
- [Background] Vera J, Ochoa J, Romero M, Vazquez-Carcano M, Ramos-Gregorio CO, Aguilar RR, Cruz A, Sleiman P, Arias A. Intracanal Cryotherapy Reduces Postoperative Pain in Teeth with Symptomatic Apical Periodontitis: A Randomized Multicenter Clinical Trial. J Endod. 2018 Jan;44(1):4-8. doi: 10.1016/j.joen.2017.08.038. Epub 2017 Nov 1. PMID 29079057
- [Derived] Ahmad MZ. Effects of intracanal cryotherapy on postoperative pain in necrotic teeth with symptomatic apical periodontitis: a randomized controlled clinical trial. Front Dent Med. 2025 Apr 14;6:1543383. doi: 10.3389/fdmed.2025.1543383. eCollection 2025. PMID 40297278